CLINICAL TRIAL: NCT05423522
Title: Prospective, Multicenter, First Part Randomized, Placebo-controlled, Parallel-group, Double-blind Period Followed by Open-label Trial Period to Evaluate Clinical Safety & Efficacy of NanoLithium® NP03 in Patients With Mild-to-severe Alzheimer's Disease: Proof-of-concept Study
Brief Title: Clinical Safety and Efficacy Evaluation of NanoLithium® NP03 in Patients With Mild-to-severe Alzheimer's Disease
Acronym: NanoLi®_AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medesis Pharma SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021 NanoLi-CT01
Record Dates: First submitted 2022-04-15; First posted 2022-06-21 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, with a first randomized, placebo-controlled, parallel-group, double-blind period followed by an open-label trial period to evaluate the clinical safety and efficacy of NanoLithium® NP03 in patients with mild-to-severe Alzheimer's disease: a proof-of-concept study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind period followed by an open-label trial period. The double-blind will be maintained throughout the double-blind period treatment (except exceptional unblinding in emergency situations for reasons of patient safety).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NanoLithium® NP03 (Experimental): Description: Homogeneous yellow oily liquid. Dosage: One administration of 3 mL per day (1.8 mg/day) by depositing 1.5 mL in the gingivo-jugal groove of each cheek with the graduated pipette.
  Duration of treatment: Approximately one year (12 weeks for the double-blind period and 36 weeks for the subsequent open-label period).
  Interventions: Drug: NanoLithium® NP03
- Placebo (Placebo Comparator): Description: Homogeneous yellow oily liquid. Dosage: One administration of 3 mL per day (1.8 mg/day) by depositing 1.5 mL in the gingivo-jugal groove of each cheek with the graduated pipette.
  Duration of treatment: 12 weeks during the double-blind period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NanoLithium® NP03 — One administration of 3 mL per day (1.8 mg/day) by depositing 1.5 mL in the gingivo-jugal groove of each cheek with the graduated pipette.
  Arms: NanoLithium® NP03
Drug: Placebo — One administration of 3 mL per day (1.8 mg/day) by depositing 1.5 mL in the gingivo-jugal groove of each cheek with the graduated pipette.
  Arms: Placebo

SUMMARY:
This proof-of-concept study will assess safety, tolerance, and efficacy of NanoLithium® NP03 in patients with mild-to-severe Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
This French Study is a prospective, multicenter, randomized (1:1), placebo-controlled, parallel-group, double-blind period followed by an open-label trial period to Evaluate Clinical Safety and Efficacy of NanoLithium® NP03 in Patients With Mild-to-severe Alzheimer's Disease.

Patients will be randomized into two treatment arms:

* NanoLithium® NP03 (N=34)
* Placebo (N=34)

The first phase will consist of a double blind 12-week -period, which will be followed by an open-label 36-week period for each arm.

A total of 18 clinical or phone call visits are scheduled during this study. During the follow-up, clinical, biological, electrophysiological, imaging assessments and questionnaires will be performed to determine the safety, efficacy, and disease-modifying effect of NanoLithium® NP03.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 50 and 90 years inclusive;
* Sufficient clinical and paraclinical information for the diagnosis of AD according to the international diagnosis criteria from McKhann G. M. et al. 2011;
* Patient presents clinically significant behavioral and psychological symptoms of dementia (BPSD) requiring medication in the opinion of the study physician (at least one item of the Neuropsychiatric Inventory-12 [NPI-12] with a score ≥ 4);
* Mild to-severe AD with a Minimal Mental State Examination (MMSE) score from 10 to 26 included;
* Symptomatic treatments of AD (acetylcholinesterase inhibitors and memantine) and psychotics drugs (benzodiazepines, antidepressants, anxiolytics, neuroleptics) are allowed but need to be maintained during at least 4 weeks before inclusion and during the follow-up;
* Female patient of childbearing potential must be willing to use an efficient birth control method during the study and until 5 days after the end of the treatment.

A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus, tubal ligation).

The following are acceptable contraceptive methods: - Established use of oral, injected, or implanted hormonal methods of contraception - Intrauterine system or placement of an intrauterine device - Double barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam, gel, film, cream, or suppository - True abstinence [periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception]

* Male patient must be willing to use male contraception (condom) during the study;
* Patient must have availability of a person ("study partner" or caregiver) who has frequent and sufficient contact with the patient, can provide accurate information regarding the patient's behavior, cognitive, and functional abilities as well as his/her health throughout the study, and agrees to provide information at investigational site visits;
* Patient is willing and able to give informed consent. If the study patient is not competent, a legally authorized representative must provide informed consent on his/her behalf, and the patient must provide assent;
* Patient affiliated to French social security;
* Patient is willing to and can comply with the study protocol requirements, in the opinion of the investigator.
* If the patient took part to another therapeutic clinical trial, he/she must systematically observe a wash-out period of > 4 weeks, or of > 6 months if he/she received a biologic disease modifying treatment (antibodies targeting the β-amyloid protein or the p-Tau protein) or 5 half-lives of investigational drug(s), whichever is longer.

Exclusion Criteria:

* Patient with genetic form of AD (known genetic mutation);
* Patient with major physical or neurosensory problems likely to interfere with the tests; contraindication or refusal to perform functional brain imaging examinations;
* Absence of caregivers to complete psychological and behavioral scales and/or questionnaires;
* Patient with illiteracy and/or inability to perform psychological and behavioral evaluations;
* Pathologies involving short term vital prognosis (progressive cancer, unstable heart failure, severe liver, kidney or respiratory diseases);
* Primary chronic psychosis or psychotic episodes not associated with the AD pathology;
* Addiction to alcohol or drugs;
* Pregnancy or breast-feeding;
* Epilepsy or other neurodegenerative disorders;
* Vitamin B12 or folic acid deficiency without supplementation;
* Patient participating in another drug trial;
* Thyroid disorders not treated;
* Patient living in institution;
* Patient deprived of liberty by law;
* Patient with contraindications to drugs containing lithium: heart failure, renal failure, Addison disease, and Brugada syndrome.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
NPI-12 total score | 12 Weeks
  The change from baseline to end of double-blind period (W12) of the NPI-12 total score in the NanoLithium® NP03 arm and in the placebo arm.

SECONDARY OUTCOMES:
Safety of treatment - Adverse effects | approximately 1 year
  The number and types of adverse effects during the study and causal role of the study treatment.
Safety of treatment - Clinical assessments - associated pathologies | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common clinical assessment: associated pathologies: medical conditions start and end date or ongoing, currently treated or not, recorded from patients file.
Safety of treatment - Clinical assessments - biochemistry - AST/ALT | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common biological tests assessment: Clinical laboratory evaluations: biochemistry: AST/ALT (UI/L)
Safety of treatment - Clinical assessments - biochemistry - Creatinine | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common biological tests assessment: Clinical laboratory evaluations: biochemistry: Creatinine (mg/L or µmol/L)
Safety of treatment - Clinical assessments - biochemistry - Glomerular filtration rate | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common biological tests assessment: Clinical laboratory evaluations: biochemistry: Glomerular filtration rate -Cockcroft or MDRD method - (ml/min/1,73m2)
Safety of treatment - Clinical assessments - biochemistry - B9 vitamin | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common biological tests assessment: Clinical laboratory evaluations: biochemistry: B9 vitamin (µg/L or nmol/L)
Safety of treatment - Clinical assessments - biochemistry - B12 vitamin | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common biological tests assessment: Clinical laboratory evaluations: biochemistry: B12 vitamin (ng/L or pmol/L)
Safety of treatment - Clinical assessments - biochemistry - T3 | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common biological tests assessment: Clinical laboratory evaluations: biochemistry: T3 (µg/L or nmol/L)
Safety of treatment - Clinical assessments - biochemistry - T4 | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common biological tests assessment: Clinical laboratory evaluations: biochemistry: T4 (µg/L or nmol/L)
Safety of treatment - Clinical assessments - biochemistry - TSH | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common biological tests assessment: Clinical laboratory evaluations: biochemistry: TSH (mlU/L)
Safety of treatment - Clinical assessments - Hematology | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common biological tests assessment: Clinical laboratory evaluations: hematology
Safety of treatment - Clinical assessments - Lithium blood level | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common biological tests assessment: Clinical laboratory evaluations: lithium blood level
Safety of treatment - Clinical assessments - Systolic and diastolic blood pressure | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common clinical assessment: Vital signs: Systolic and diastolic blood pressure (mm Hg)
Safety of treatment - Clinical assessments - Pulse rate | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common clinical assessment: Vital signs: Pulse rate (beats per minute [bpm])
Safety of treatment - Clinical assessments - ECG - PR | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common clinical assessment: Electrocardiogram (ECG): PR interval (msec)
Safety of treatment - Clinical assessments - ECG - QRS | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common clinical assessment: Electrocardiogram (ECG): QRS interval (msec)
Safety of treatment - Clinical assessments - ECG - QT | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common clinical assessment: Electrocardiogram (ECG): QT interval (msec)
Safety of treatment - Clinical assessments - ECG - RR | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common clinical assessment: Electrocardiogram (ECG): RR interval (msec)
Safety of treatment - Clinical assessments - ECG - QTcB | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common clinical assessment: Electrocardiogram (ECG): QTcB interval (msec)
Safety of treatment - Clinical assessments - Weight | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common clinical assessment: General clinical examination: weight (in Kg)
Safety of treatment - Clinical assessments - Height | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common clinical assessment: General clinical examination: height (in cm)
Safety of treatment - Clinical assessments - BMI | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common clinical assessment: General clinical examination: body mass index (BMI) (weight and height will be combined to report BMI in kg/m^2)
Safety of treatment - Clinical assessments - cognitive signs | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common neurological assessments: Neurological clinical examination: cognitive signs: questions asked to patients/caregiver to detect execution troubles, attention troubles, language, gnosic troubles, praxis, visuo-spacial troubles and temporo-spacial orientation
Safety of treatment - Clinical assessments - focal neurological signs | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common neurological assessments: Neurological clinical examination: focal neurological signs: questions asked to patients/caregiver to detect extrapyramidal syndrome, pyramidal syndrome, cerebellar syndrome, frontal syndrome, hallucinations, dysautonomia, sensitive system and epilepsy
Safety of treatment - Clinical assessments - motricity | approximately 1 year
  To assess the safety of NanoLithium® NP03 after 48 weeks of treatment based on common neurological assessments: Neurological clinical examination: motricity: questions asked to patients/caregiver to detect muscular tonus, abnormal movements, reflex, walking troubles, falls, postural troubles, coordination, sphincter and trophic troubles
Efficacy of treatment_BPSD_NPI-C-IPA | After 12 and 48 weeks
  To assess the BPSD at 12 and 48 weeks, change from baseline to week 12 and week 48 on the Neuropsychiatric Inventory - Clinician items mapped to International Psychogeriatric Association (NPI-C-IPA) scale (Units on a Scale).
Efficacy of treatment_BPSD_NPI-12 | After 12 and 48 weeks
  To assess the BPSD at 12 and 48 weeks, score of each item of the Neuropsychiatric Inventory (NPI-12) (Units on a Scale).
Efficacy of treatment_cognitive performances - MMSE Score | After 12 and 48 weeks
  MMSE score (Units on a Scale).
Efficacy of treatment_cognitive performances - CDRS Score | After 12 and 48 weeks
  Clinical Dementia Rating Scale (CDRS) score (Units on a Scale).
Efficacy of treatment_cognitive performances - ADL Score | After 12 and 48 weeks
  Activity of Daily Living (ADL) score (Units on a Scale).
Efficacy of treatment_PET-FDG | After 12 and 48 weeks
  Cerebral metabolic rate for glucose measured by Positron Emission Tomography-Fluorodeoxyglucose (PET-FDG).
Efficacy of treatment_Biomarkers_Peripheral biomarkers | After 12 and 48 weeks
  Pathophysiological peripheral biomarkers (amyloid biomarkers, neurofilaments, Tau protein, BDNF) (pg/ml).
Efficacy of treatment_Biomarkers_Non-specific biomarkers | After 12 and 48 weeks
  Non-specific biomarkers (inflammation cytokines).
Efficacy of treatment_Drug compliance | After 12 and 48 weeks
  Drug compliance by assessing the number of buccal deposits.

CONTACTS AND LOCATIONS:
Overall Officials: Maria SOTO MARTIN, Prof., Principal Investigator — CHU Toulouse - Hôpital La Grave - Cité de la Santé
Locations (8):
- France (8):
  - CHU de Lille, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Hôpital De La Timone, Marseille
  - CHU de Montpellier - Hôpital Gui de Chauliac, Montpellier
  - Hôpital Lariboisière, Paris
  - Hôpital Universitaire de Strasbourg, Strasbourg
  - CHU Toulouse - Hôpital La Grave - Cité de la Santé, Toulouse
  - Hôpital des Charpennes - Hospices Civils de Lyon, Villeurbanne